CLINICAL TRIAL: NCT03979508
Title: Window Trial of Abemaciclib for Surgically Resectable, Chemotherapy-Resistant, Triple Negative Breast Cancer (a BEAUTY Study*)
Brief Title: Abemaciclib in Treating Patients With Surgically Resectable, Chemotherapy Resistant, Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary biomarker (CD8/FOXP3) was rarely observed to be < 1.6 in residual tumors examined in first stage of study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1734; NCI-2019-03567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1734 (Other: Mayo Clinic in Rochester); 17-010660 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Breast Ductal Carcinoma In Situ; Breast Fibrocystic Change; Breast Lobular Carcinoma In Situ; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Fibrocystic Breast Disease; Breast Carcinoma In Situ; Triple Negative Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A Group 1; Cohort B Group 3 (surgery) (Experimental): Patients undergo standard of care surgical resection.
  Interventions: Procedure: Therapeutic Conventional Surgery
- Cohort A Group 2; Cohort B Group 4 (abemaciclib, surgery) (Experimental): Patients receive abemaciclib PO BID on days 1-14 or days 1-21 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgical resection no later than 12 weeks after the last dose of neoadjuvant chemotherapy.
  Interventions: Drug: Abemaciclib; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
  Arms: Cohort A Group 2; Cohort B Group 4 (abemaciclib, surgery)
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgical resection

SUMMARY:
This phase II trial studies how well abemaciclib works in treating patients with triple negative breast cancer that can be removed by surgery (resectable) and does not respond to treatment with chemotherapy alone, or in combination with pembrolizumab. Abemaciclib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the effects of abemaciclib on the CD8/FOXP3 ratio in chemotherapy resistant triple negative breast cancer (TNBC) patients following neoadjuvant chemotherapy regimen without the addition of pembrolizumab (Cohort A).

II. To examine the effects of abemaciclib on the CD8/FOXP3 ratio in chemotherapy resistant TNBC patients following a neoadjuvant chemotherapy regimen with the addition of pembrolizumab (Cohort B).

SECONDARY OBJECTIVES for Cohort A and Cohort B Independently:

I. Assess abemaciclib toxicities. II. To examine the effects of abemaciclib on the percentage of vimentin expressing invasive cancer cells

III. Within TNBC molecular subtypes (basal, mesenchymal, and luminal androgen receptor [LAR]), to evaluate the effects of abemaciclib on:

IIIa. The individual elements of tumor grade (mitoses, nuclear pleomorphism, and tubule formation).

IIIb. Tumor proliferation (as measured by tumor Ki-67 and serum tyrosine kinase inhibitor [TKI]).

IIIc. pDUB3 as well as epithelial-mesenchymal transition (EMT) markers including SNAIL/SLUG, TWIST, and E-Cadherin as measured by immunohistochemistry (IHC).

IIId. Quantification of tumor-infiltrating lymphocytes (as examined by hematoxylin and eosin [H&E]).

EXPLORATORY OBJECTIVES for Cohort A and Cohort B Independently:

I. To evaluate the effect of abemaciclib on tumor ribonucleic acid (RNA) expression.

II. To evaluate the effects of abemaciclib on the immune phenotype of peripheral blood mononuclear cells (PBMC), by evaluating expression of a panel of cell surface markers optimized of identification of human immune cell subpopulations.

III. To evaluate the effects of abemaciclib on tumor-infiltrating immune cells in formalin-fixed paraffin-embedded (FFPE) tumor sections, using multiplexed imaging technologies (e.g imaging mass cytometry, Nanostring digital spatial profiling [DSP] or CODEX) which will include:

IIIa. Genes directly involved in tumor cell antigen presentation (e.g. B2M, HLA-A, HLA-B, HLA-C, TAP1, TAP2, TAPBP).

IIIb. Interferon-stimulated genes (ISGs) that regulate antigen presentation (e.g. STAT1, NLRC5) and other ISGs (e.g. IRFs, OAS2).

IIIc. Genes involved in double-strand ribonucleic acid (dsRNA) response (e.g. DDX58, DHX58).

IIId. Genes encoding interferons, including type 3 IFNs (e.g. IFNL1, IFNL2, IFNL3).

IIIe. Genes indicating a cytotoxic T cell response (e.g. PRF1, GZMB). IIIf. Regulatory T-cell (Treg)-specific transcription factor genes (e.g. FOXP3, IKZF2).

IV. To assess the difference in the frequency of JAK-2 amplification among patients whose post-abemaciclib CD8/FOXP3 ratio >= 1.6 and that among patients whose post-abemaciclib CD8/FOXP3 ratio < 1.6.

V. To generate organoids for future research. VI. To evaluate changes in the microbiome with exposure to abemaciclib.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT A: Patients receive a neoadjuvant chemotherapy regimen without pembrolizumab.

GROUP 1: Patients undergo standard of care surgical resection.

GROUP 2: Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-14 or days 1-21 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgical resection no later than 12 weeks after the last dose of neoadjuvant chemotherapy.

After completion of study treatment, patients in group 2 are followed up within 30-60 days.

COHORT B: Patients receive a neoadjuvant chemotherapy regimen in combination with pembrolizumab.

GROUP 3: Patients undergo standard of care surgical resection.

GROUP 4: Patients receive abemaciclib orally (PO) twice daily (BID) on days 1-14 or days 1-21 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care surgical resection no later than 12 weeks after the last dose of neoadjuvant chemotherapy.

After completion of study treatment, patients in group 4 are followed up within 30-60 days.

ELIGIBILITY:
Inclusion Criteria:

* Women of age >=18 years
* PRE-REGISTRATION: Clinical T1-4, N0-3, M0 breast cancer at diagnosis (prior to the start of neoadjuvant chemotherapy) by American Joint Committee on Cancer (AJCC) staging version 8.

  * Note: Benign breast disease, lobular carcinoma in situ (LCIS) or ductal carcinoma in situ (DCIS) in the ipsilateral or contralateral breast is allowed.
  * Note: Additional ipsilateral or contralateral invasive breast cancer is allowed. The index lesion is the largest triple-negative, chemotherapy-resistant lesion.
* PRE-REGISTRATION: Histological confirmation of triple negative invasive breast cancer (defined as estrogen receptor [ER] =< 10%, progesterone receptor [PR] =< 10% and HER2 not amplified by in situ hybridization [ISH] or immunohistochemistry [IHC] 0/1) at diagnosis.
* PRE-REGISTRATION: Cohort A: CLOSED TO PRE-REGISTRATION and REGISTRATION as of protocol amendment 6 (04/14/2023) Neoadjuvant chemotherapy (NAC) with one of the following regimens that was not discontinued early due to intolerability with less than 50% of planned treatment given due to disease progression or patient request:

  * Paclitaxel or docetaxel followed by one of the following: the combination of doxorubicin and cyclophosphamide (AC); the combination of epirubicin and cyclophosphamide (EC) or the combination of 5-fluorouracil, epirubicin and cyclophosphamide (FEC)

    * Note: Carboplatin may be added to these regimens
  * AC or EC or FEC followed by docetaxel or paclitaxel

    * Note: Carboplatin may be added to these regimens
  * Docetaxel in combination with doxorubicin and cyclophosphamide (TAC)
  * Docetaxel in combination with cyclophosphamide (TC) (for patients who are not candidates for anthracyclines)
  * Carboplatin or cisplatin in combination with a taxane (paclitaxel, docetaxel, or nab-paclitaxel) (for patients who are not candidates for anthracyclines)
* PRE-REGISTRATION: Cohort B: Neoadjuvant chemotherapy (NAC) with one of the following regimens in combination with pembrolizumab that was not discontinued early due to intolerability with less than 50% of planned treatment given due to disease progression or patient request:

  * Paclitaxel or docetaxel followed by one of the following: the combination of doxorubicin and cyclophosphamide (AC); the combination of epirubicin and cyclophosphamide (EC) or the combination of 5-fluorouracil, epirubicin and cyclophosphamide (FEC) Note: Carboplatin may be added to these regimens
  * AC or EC or FEC followed by docetaxel or paclitaxel [Note: Carboplatin may be added to these regimens]
  * Docetaxel in combination with doxorubicin and cyclophosphamide (TAC)
  * Docetaxel in combination with cyclophosphamide (TC)
  * Carboplatin or cisplatin in combination with a taxane (paclitaxel, docetaxel, or nab-paclitaxel)
* PRE-REGISTRATION: Residual lesion/enhancement seen in the breast on breast imaging performed after completion of NAC.
* PRE-REGISTRATION: Able to swallow oral medication.
* PRE-REGISTRATION: Willing to undergo biopsy for research.
* PRE-REGISTRATION: Willing to provide tissue and blood samples for correlative research purposes.
* PRE-REGISTRATION: Willing to stop use of strong and moderate inducers and/or strong inhibitors of cytochrome P450 3A =< 7 days prior to registration.
* PRE-REGISTRATION: Provide written informed consent.
* REGISTRATION: Registration must occur =< 56 days after last dose of NAC.
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2.
* REGISTRATION: COHORT B GROUP 4 ONLY: The following laboratory values obtained after completion of NAC but =< 14 days prior to registration:
* REGISTRATION: COHORT B GROUP 4 ONLY: Absolute neutrophil count (ANC) >= 1500/mm^3.
* REGISTRATION: COHORT B GROUP 4 ONLY: Platelets (PLT) >= 100,000/mm^3.
* REGISTRATION: COHORT B GROUP 4 ONLY: Hemoglobin (HgB) >= 8.0 g/dL.
* REGISTRATION: COHORT B GROUP 4 ONLY: Total bilirubin =< 1.5 x upper limit of normal (ULN).
* REGISTRATION: COHORT B GROUP 4 ONLY: Aspartate transaminase (AST) serum glutamic oxaloacetic transaminase (SGOT) =< 3 x ULN.
* REGISTRATION: COHORT B GROUP 4 ONLY: Alanine transaminase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 3 x ULN.
* REGISTRATION: COHORT B GROUP 4 ONLY: Serum creatinine =< 1.5 x ULN.
* REGISTRATION: GROUP 2 ONLY: Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only.

Exclusion Criteria:

* PRE-REGISTRATION: History of deep venous thrombosis (DVT) or pulmonary embolisms (PE) =< 12 months prior to preregistration; OR Active DVT and/or PE requiring anti-coagulant therapy.

  * NOTE: Patients who are on anti-coagulant therapy for maintenance are eligible as long as the DVT and/or PE was > 12 months prior to enrollment and there is no evidence for active thrombosis (either DVT or PE).
  * NOTE: Patients on anticoagulation are eligible; however peri-biopsy and peri-surgical management of anticoagulation is per the institutional standard of care.
* PRE-REGISTRATION: Prior treatment with CDK 4/6 inhibitors (e.g. palbociclib, ribociclib, abemaciclib, etc.)
* PRE-REGISTRATION: Prior treatment with radiation for this breast cancer.
* PRE-REGISTRATION: Prior incisional or excisional breast biopsy for this cancer.
* PRE-REGISTRATION: Any contraindications to pre-registration biopsy (such as bleeding diatheses, etc.).
* PRE-REGISTRATION: Receiving any investigational agent which would be considered as a treatment for the primary neoplasm.
* PRE-REGISTRATION: Other active malignancy =< 3 years prior to registration.

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix.
  * NOTE: If there is a history of prior malignancy, they must not be receiving another specific treatment for prior malignancy.
* PRE-REGISTRATION: Biopsy proven Stage IV breast cancer.
* PRE-REGISTRATION: Serious pre-existing medical conditions that would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g., estimated creatinine clearance < 30 ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline grade 2 or higher diarrhea).
* PRE-REGISTRATION: History of any of the following conditions:

  * Syncope of cardiovascular etiology.
  * Ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation).
  * Sudden cardiac arrest.
  * NOTE: Patients on anticoagulation are eligible; however peri-biopsy and peri-surgical management of anticoagulation is per the institutional standard of care.
* REGISTRATION: COHORT B GROUP 4: Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons.
  * Nursing persons.
  * Persons of childbearing potential who are unwilling to employ adequate contraception.
* REGISTRATION: COHORT B GROUP 4: Failure to recover to grade 1 or lower from effects of neoadjuvant chemotherapy.

  * Exceptions: Residual alopecia and grade 2 peripheral neuropathy are allowed.
* REGISTRATION: COHORT B GROUP 4: Concurrent use of strong and moderate inducers and/or strong inhibitors of cytochrome P450 3A =< 7 days prior to registration.
* REGISTRATION: COHORT B GROUP 4: Known infections as follows (NOTE: Screening is not required for enrollment):

  * Active systemic bacterial infection requiring intravenous antibiotics.
  * Active fungal infection (requiring intravenous or oral antifungal treatment).
  * Detectable viral infections (e.g. known human immunodeficiency virus [HIV], known active hepatitis B or C).
* REGISTRATION: COHORT B GROUP 4: Concurrent use of chemotherapy, radiotherapy, immunotherapy, or other components of neoadjuvant treatment.

  * NOTE: Patients must complete all elements of NAC ≥21 days prior to starting abemaciclib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have a CD8/FOXP3 ratio < 1.6 in their residual tumors after neoadjuvant chemotherapy (NAC) that convert to CD8/FOXP3 ratio >= 1.6 | Up to 21 days
  A Simon optimum two stage phase II clinical trial design was chosen to test the null hypothesis that the rate of conversion to post-abemaciclib CD8/FOXP3 ratio of 1.6 or more is =< 5% against the alternative that rate of conversion to post-abemaciclib CD8/FOXP3 ratio of 1.6 or more is >= 20% with the target probability of a type I error and probability of a type II error set to 0.10. The probability of terminating after the first stage is 0.736, if the null hypothesis is true. A 90% confidence interval for this rate of conversion will be constructed using the Duffy-Santner approach taking into account the sequential nature of the study

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 60 days
  Adverse events will be monitored and graded with attribution assigned using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. For each type of adverse event (AE) reported, the proportion of patients experiencing a grade 2 or worse level of that AE will be determined.
Changes in vimentin expression | Up to 60 days
  Vimentin expression will be evaluated by immunohistochemistry (IHC) with using 0, 1+, 2+ or 3+ scoring scheme. A point estimate of the proportion of eligible patients whose post-NAC residual tumor Vimentin expression levels were 2+ or 3+ and then fell to 0 or 1+ after abemaciclib among the eligible patients whose began abemaciclib treatment after a post NAC residual tumor Vimentin expression level finding of 2+ or 3+ will be calculated. A 90% confidence interval for this proportion will be constructed using one-sample binomial confidence for proportions.
Impact of length of treatment | Up to 60 days
  Association between amount of abemaciclib received and the change in CD8/FOXP3 ratio after abemaciclib will be explored graphically. A plot of the change in change in CD8/FOXP3 ratio after abemaciclib and days of treatment will be constructed to visually assess for trends. Also, the a 90% confidence interval for the difference in binomial proportions will be constructed to assess whether the proportion of patients whose post abemaciclib CD8/FOXP3 ratio >= 1.6 after completing 14-21 days of abemaciclib differs between those who discontinued abemaciclib the day prior to surgery and who discontinued abemaciclib 2 or more days prior to surgery. A 90% binomial confidence interval for the proportion of women who failed to complete 14-21 days of abemaciclib or underwent surgery or breast biopsy 2 or more days after last dose of abemaciclib among the eligible women who began abemaciclib treatment.

OTHER OUTCOMES:
Changes in mitoses | Up to 60 days
  Examined graphically overall and by triple negative breast cancer (TNBC) subtypes.
Changes in nuclear pleomorphism | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in tubule formation | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in tumor Ki-67 | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in serum tyrosine kinase inhibitor (TKI) | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in SNAIL | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in SLUG | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in E-Cadherin | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Changes in tumor-infiltrating lymphocytes | Up to 60 days
  Examined graphically overall and by TNBC subtypes.
Effect of abemaciclib on tumor ribonucleic acid (RNA)-sequencing (seq) data | Up to 60 days
  Effect of abemaciclib on tumor RNA sequencing followed by standard and customized pathway and enrichment analysis (e.g., Gene set enrichment analysis (GSEA) and CIBERSORT methods). The GSEA method determines whether an a priori set of genes are over-represented in the differential expression analysis of the pre- and post- drug response phenotypes. Similarly, CIBERSORT estimates cell composition from RNA transcriptomic data (e.g. immune cell populations).
Effect of abemaciclib on the phenotype of peripheral blood mononuclear cells (PBMC) | Up to 60 days
  Will be assessed using mass cytometry (e.g,. CyTOF) to analyze a panel of 29 cell surface markers optimized for identification of human immune cell subsets, including the following targets: CD45, CD195 (CCR6), CD19, CD127, CD38, IgD, CD11c, CD16, CD194 (CCR4), CD123/IL-3R, TCRgd, CD185 (CXCR5), CD3, CD45RA, CD27, CD29, CD66b, CD183 (CXCR3), CD161, CD45RO, CD197 (CCR7), CD8a, CD25/IL-2R, CD20, HLA-DR, CD4, CD14, CD56/NCAM. Identification of specific immune cell subsets will be assessed using consensus clustering methods of predefined combination of markers.
Effect of abemaciclib on formalin-fixed paraffin-embedded (FFPE) tumor sections | Up to 60 days
  Will include (imaging mass cytometry multiplex quantitative RNA/protein immune-based profilings, such as Hyperion TM, Nanostring GeoMX, Codex, and may include the examination of genes directly involved in tumor cell antigen presentation (e.g. B2M, HLA-A, HLA-B, HLA-C, TAP1, TAP2, TAPBP), interferon-stimulated genes (ISGs) that regulate antigen presentation (e.g. STAT1, NLRC5) and other ISGs (e.g. IRFs, OAS2), genes involved in double strand RNA response (e.g. DDX58, DHX58), genes encoding interferons, including type 3 IFNs (e.g. IFNL1, IFNL2, IFNL3), genes indicating a cytotoxic T cell response (e.g. PRF1, GZMB), regulatory T cell-specific transcription factor genes (e.g., FOXP3, IKZF2)
Change in in frequency of JAK-2 amplifications | Baseline up to time of surgery
  The collection of JAK-2 will be used to assess the difference in the frequency of JAK-2 amplification among patients whose post-abemaciclib CD8/FOXP3 ratio >= 1.6 and that among patients whose post-abemaciclib CD8/FOXP3 ratio < 1.6. A 95% binomial confidence for the difference in two independent proportions will be constructed for the difference in the percentage of patients with a post-abemaciclib CD8/FOXP3 ratio >= 1.6 among those with JAK-2 amplified TNBC and those with JAK-2 non-amplified TNBC.
Change in microbiome with exposure to abemaciclib | Baseline up to prior to surgery
  The collection of microbiome information via stool collection will be used to generate descriptive analyses about the study population, as the total number of samples is expected to be insufficient for full statistical analysis. Will explore putative mechanistic connections underlying bacteria-drug interactions in all patients and attempt to identify the biomolecular features within the gut (stool) microbiome and its association with the pharmacokinetics and pharmacodynamics of abemaciclib.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P. Goetz, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03979508/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT03979508/ICF_001.pdf